CLINICAL TRIAL: NCT05824338
Title: Testing the Feasibility of Using Ropivacaine in Spinal Anesthesia for Patients With Lower Back Surgery
Acronym: SASS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fraser Health (Other)
Responsible Party: Principal Investigator, Alan Tung, Clinical Instructor, Fraser Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022430
Record Dates: First submitted 2023-03-09; First posted 2023-04-21 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia, Spinal; Neurosurgery; Ropivacaine; Bupivacaine
Keywords: Anesthesia; Spinal; Lumbar surgery; Lower back
MeSH Terms: interventions — Anesthesia, Spinal; Ropivacaine; Bupivacaine; Anesthesia, General; Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General anesthesia with endotracheal tube (Active Comparator): Currently the standard at our centre. Participants in this group will undergo lower lumbar surgery with general anesthesia with endotracheal intubation.
  Interventions: Drug: General anesthesia for lumbar surgery
- Spinal anesthesia with bupivacaine (Active Comparator): Participants in this group will undergo lower lumbar surgery under spinal anesthesia with bupivacaine 0.5% 10-15 mg with fentanyl 10-15 mcg.
  Interventions: Drug: Spinal anesthesia for lumbar surgery: bupivacaine
- Spinal anesthesia with ropivacaine (Experimental): Participants in this group will undergo lower lumbar surgery under spinal anesthesia with ropivacaine 0.5% 10-20 mg with fentanyl 10-15 mcg.
  Interventions: Drug: Spinal anesthesia for lumbar surgery: ropivacaine

INTERVENTIONS:
Drug: Spinal anesthesia for lumbar surgery: ropivacaine — The anesthesiologist will administer 4 mL of ropivacaine 0.5% plus fentanyl 15 mcg intrathecally
  Other Names: Ropivacaine in the spinal anesthesia for lower lumbar surgery
  Arms: Spinal anesthesia with ropivacaine
Drug: Spinal anesthesia for lumbar surgery: bupivacaine — The anesthesiologist will administer 3 mL of bupivacaine 0.5% plus fentanyl 15 mcg intrathecally.
  Other Names: Bupivacaine in the spinal anesthesia for lower lumbar surgery
  Arms: Spinal anesthesia with bupivacaine
Drug: General anesthesia for lumbar surgery — Patient will be intubated and ventilated under general anesthesia.
  Other Names: General Anesthesia with Endotracheal intubation
  Arms: General anesthesia with endotracheal tube

SUMMARY:
The goal of this pilot clinical trial is to test the feasibility of conducting a randomized controlled trial that will examine the use of ropivacaine in the spinal anesthesia for patients undergoing elective 1- or 2-level lower spine surgery. This study aims to:

* Determine the rates of eligibility, recruitment, consent, and attrition
* Determine the acceptability among patients, surgeons, anesthesiologists, and nurses of doing spine surgery under spinal anesthesia
* Gather preliminary data on outcomes relevant to a future dose-finding study

Participants will be randomized to one of three treatment groups:

* General anesthesia with endotracheal tube
* Spinal anesthesia with bupivacaine
* Spinal anesthesia with ropivacaine

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are equal to or greater than 18 years old
* Undergoing elective one or two-level lumbar surgery via posterior surgical approach in the prone position (between L2-S1)
* Expected surgery duration of no greater than 2 hours
* ASA Physical Status Class 1 to 3
* Patient can have either spinal anesthesia or general anesthesia
* Able to provide consent and understand information in English, and capable of answering questions in English

Exclusion Criteria:

* Allergy to either ropivacaine, bupivacaine, or local anesthetics
* Contraindications to spinal anesthesia (i.e. coagulopathy or on anticoagulants, severe aortic or mitral valve stenosis, sepsis or bacteremia, thrombocytopenia, high intracranial pressure, infection at the puncture site)
* Surgery is expected to take more than 2 hours
* Emergency surgery
* Previously had back surgery at the level of the spine currently being operated on
* Comorbidities that require the patient to undergo general anesthesia
* Inability to stay still during the surgery
* Inability to move legs preoperatively
* Body Mass Index (BMI) >35
* Multilevel severe spinal stenosis

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of study procedures and intervention: eligibility and recruitment | Study duration, until last patient has completed the study (average of 1 year)
  Number of patients contacted who accepted or declined to participate in the study, with the acceptance rate calculated as the percentage of contacted patients who agreed to participate in the study
Acceptability of study procedures and intervention: attrition | Study duration, until last patient has completed the study (average of 1 year)
  Number of patients who complete the study after randomization, with the completion rate calculated as the percentage of randomized patients in whom we were able to collect the Quality of Recovery-15 survey results
Acceptability of study procedures and intervention: attrition (reasons) | Study duration, until last patient has completed the study (average of 1 year)
  Reasons why the patient, neurosurgeon and/or anesthesiologist refused to proceed with the patient's pilot study participation
Determining the success of our randomization procedures: as per protocol | Study duration, until last patient has completed the study (average of 1 year)
  Number of participants who actually get the intervention assigned to them, calculated as the percentage of randomized patients who receive the anesthetic protocol assigned to them
Determining the success of our randomization procedures: randomization process | Study duration, until last patient has completed the study (average of 1 year)
  Similarity of the groups on their baseline characteristics based on the demographic information

SECONDARY OUTCOMES:
Preliminary outcome data: height of sensory block after intrathecal administration of study medications | Intraoperative and postoperative up to 24 hours (per patient); study duration after last patient has completed the study (average of 1 year)
  Assessing for dermatome level at which the patient has normal sensation to ice and pinprick, at specific intervals (every 2 minutes after spinal anesthesia up to 10 minutes or until thoracic level between T10 and T6 is achieved (whichever is later); on arrival to PACU; every 30 minutes after arrival to PACU until discharge to the ward or home).
Preliminary outcome data: density of sensory block after intrathecal administration of study medications | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  whether the patient is able to sense nothing, touch, or pain at time of first incision
Preliminary outcome data: motor block after intrathecal administration of study medications | Intraoperative and postoperative up to discharge (per patient); study duration after last patient has completed the study (average of 1 year)
  assess for muscle strength at specific intervals (every 5 minutes up to 10 to 20 minutes after spinal anesthesia, on arrival to PACU (postanesthetic recovery unit), and every 30 minutes after arrival to PACU until discharge to the ward or home).
Preliminary outcome data: pain scores | Intraoperative and postoperative up to 24 hours (per patient); study duration after last patient has completed the study (average of 1 year)
  preoperatively; intraoperatively; on arrival to PACU (postanesthetic recovery unit); at discharge from PACU to the ward or home; 24 hours after surgery. Measure: numerical rating scale (0 to 10, with 10 being excruciating pain)
Preliminary outcome data: total dosages of analgesics and sedatives ( | Intraoperative and postoperative up to 24 hours (per patient); study duration after last patient has completed the study (average of 1 year)
  Total dosage of opioids and other analgesics (i.e., acetaminophen, NSAIDs) administered to the participant during surgery, and over 24 hours after surgery, as measured using milligrams
Preliminary outcome data: hypotension | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  total duration of time (in minutes) with mean arterial pressure (MAP) below 65
Preliminary outcome data: bradycardia | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  total duration of time (in minutes) with heart rate below 55
Preliminary outcome data: vasopressor requirements | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  total dose of vasopressors used intraoperatively, as measured in milligrams
Preliminary outcome data: completion rate | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Percentage of participants in the spinal anesthesia group who successfully complete their lower back surgery without additional interventions (including conversion from spinal anesthesia to general anesthesia, additional analgesics through the intravenous line, additional spinal anesthesia medication dose given by the neurosurgeon, additional numbing medication infiltrated in the surgical incision by the neurosurgeon)
Preliminary outcome data: surgery abandonment rate | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  by the number of patients who had spinal anesthesia who then had to be converted to general anesthesia or not complete surgery
Preliminary outcome data: time | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  As measured in minutes, the time it takes to: from entering the operating room to the receiving the general anesthesia or spinal anesthesia medication, to the participant being in surgical position (lying on his/her stomach), to achieve sensory level of dermatomal level between T10 and T6 (numbness to ice and pinprick)
Preliminary outcome data: neurosurgeon's experience with conducting neurosurgery under neuraxial technique, and reasons | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Whether the neurosurgeon found operating on the spine to be more or less challenging under spinal anesthesia, in comparison to his or her previous experience with general anesthesia. This will be measured on a 5-point Likert scale, from "significantly less challenging" to "significantly more challenging".
Preliminary outcome data: neurosurgeon's experience with conducting neurosurgery under neuraxial technique | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Whether the neurosurgeons would recommend doing lumbar spine surgery under spinal anesthesia as a feasible anesthetic option, measured on a 5-point Likert scale (from "very likely" to "very unlikely")
Preliminary outcome data: operating room nurses' experience with conducting neurosurgery under neuraxial technique | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Whether the operating room nurses would recommend doing lumbar spine surgery under spinal anesthesia as a feasible anesthetic option, measured on a 5-point Likert scale (from "very likely" to "very unlikely")
Preliminary outcome data: operating room nurses' workload experience with conducting neurosurgery under neuraxial technique | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Operating room nurses' workload when helping with a spine surgery conducted under spinal anesthesia, compare to when helping with a spine surgery done under general anesthesia. . This would be measured on a 5-point Likert scale, from "significantly less work (compared to GA)" to "significantly more work (compared to GA)"
Preliminary outcome data: postanesthetic care unit (PACU) nurses' experience | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Whether the PACU nurses would recommend having lumbar spine surgery done under spinal anesthesia as a feasible anesthetic option, measured on a 5-point Likert scale (from "very likely" to "very unlikely")
Preliminary outcome data: postanesthetic care unit (PACU) nurses' workload experience with conducting neurosurgery under neuraxial technique | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Postanesthetic care unit nurse (PACU) nurses' workload when taking care of a patient post-operatively from a spine surgery done under spinal anesthesia, compared to if the spine surgery had been done under general anesthesia. This would be measured on a 5-point Likert scale, from "significantly less work (compared to GA)" to "significantly more work (compared to GA)".
Preliminary outcome data: number of attempts for the anesthesiologist to administer intrathecal medications | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Graded as 1 attempt, 2 attempts, ≥3 attempts, abandoned attempt, or no attempt made (i.e. general anesthesia).
Preliminary outcome data: anesthesiologist's workload when conducting neurosurgery under spinal anesthesia | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Anesthesiologists' workload when doing the spine surgery under spinal anesthesia, in comparison to general anesthesia. This would be measured on a 5-point Likert scale, from "significantly less work (compared to GA)" to "significantly more work (compared to GA)".
Preliminary outcome data: patient's experience during spinal anesthesia administration | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Patients' experience during the administration of spinal anesthesia (inserting a needle into the back) in terms of pain tolerability. This will be assessed using the numerical rating scale (NRS). The NRS is a clinically used, validated scoring system ranging from 0 (no pain) to 10 (severe, excruciating pain
Preliminary outcome data: patient's comfort during surgery | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Patients' comfort during the surgery if they received a spinal anesthetic. This will be assessed using the NRS (described above). There will also be 2 other options to choose from in case the patient is unable to report the pain level using the numerical rating scale (NRS), including "Patient does not remember", and "N/A (patient was in general anesthesia group)".
Preliminary outcome data: patient's memory during surgery | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Whether patients who had spinal anesthesia remembered what happened during surgery. There will be 2 options: "Yes, I remember", and "No, I do not remember".
Preliminary outcome data: patient's discomfort with numbness or weakness postoperatively | Postoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  For patients who had spinal anesthesia, they are asked whether they were bothered by the weakness and/or numbness in the legs in the PACU
Preliminary outcome data: patient's preference preoperatively | Preoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  The patients are asked if, prior to surgery, they had a preference for general anesthesia or spinal anesthesia. There will be three options: "I would prefer general anesthesia", "I would prefer spinal anesthesia", and "I have no preference".
Preliminary outcome data: patient's Quality of Recovery (QoR-15) | Postoperative (per patient); study duration after last patient has completed the study (24 hours after surgery) (average of 1 year)
  QoR-15 (Quality of Recovery) score, done 24 hours after surgery, covers a range of items including ease of breathing, enjoyment of food, feeling rested, sleep quality, able to do personal hygiene unaided, communication with friends and family, able to return to work and usual home activities, feeling of being in control, overall general well-being, pain levels, nausea or vomiting, anxiety, and depression. It is scored out of 150, with a higher score signifying better quality of recovery.

OTHER OUTCOMES:
Assessing appropriateness of data collection intervals | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Whether assessing the sensory and motor blocks by 10 to 20 minutes after spinal anesthesia is long enough to determine whether the spinal anesthesia dose has achieved a minimum sensory level to dermatomal level between T10 and T6 to ice and pinprick. We will thus be monitoring the time it takes to achieve this level (measured in minutes) as noted above.
Incidence of complications from spinal anesthesia: anemia | Intraoperative and postoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Drop in hemoglobin will be measured as a percentage in hemoglobin drop, as calculated by the preoperative hemoglobin minus the postoperative hemoglobin on postoperative day 1, then divided by the preoperative hemoglobin
Incidence of intraoperative complications from spinal anesthesia | Intraoperative (per patient); study duration after last patient has completed the study (average of 1 year)
  Aggregate of complications (percentage of patients) who had issues during surgery (estimated blood loss (millilitres), incidence of low blood pressure (mean arterial pressure less than 65), incidence of low heart rate (less than 55), incidence of interventions to treat low blood pressure and/or low heart rate)
Incidence of postoperative complications from spinal anesthesia | Postoperative up to 24 hours (per patient); study duration after last patient has completed the study (average of 1 year)
  Incidence of common side effects at 24 hours after surgery from spinal anesthesia or general anesthesia, including headache, nausea, vomiting, pruritus, dizziness, blurred vision, urinary retention, numbness or tingling in the upper extremities, sore throat, as well as any other side effects not mentioned
Incidence of other postoperative complications | Postoperative up to 24 hours (per patient); study duration after last patient has completed the study (average of 1 year)
  Incidence of complications after surgery and up to discharge from hospital (headache after surgery, delirium or confusion, urinary retention requiring a Foley bladder catheter, need to return to the operating room for emergency re-operation, spinal hematoma, worsening nerve injury).
Incidence of other postoperative complications: neurological symptoms | Postoperative up to 24 hours (per patient); study duration after last patient has completed the study (average of 1 year)
  Worsening in neurological symptoms at 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alan Tung, MD, Principal Investigator — Anesthesiologist
Locations (2):
- Canada (2):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Eagle Ridge Hospital, Port Moody, British Columbia

IPD SHARING:
Plan to Share IPD: No